CLINICAL TRIAL: NCT04413708
Title: Novel mHealth Technologies to Enhance PrEP Adherence Among Thai MSM: Collaborative Adaptation and Evaluation
Brief Title: mHealth Technologies to Enhance PrEP Adherence Among Thai MSM
Acronym: P3-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Chulalongkorn University (Other); Thai Red Cross AIDS Research Centre (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-0099; 1R21TW010965 (NIH)
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Adherence, Patient; Pre-Exposure Prophylaxis; HIV/AIDS
Keywords: PrEP adherence; HIV; Young men who have sex with men; YMSM; Thailand; Mobile app; mHealth
MeSH Terms: conditions — Patient Compliance; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Model Description Definition: Provide details about the Interventional Study Model. Limit: 1000 characters.
Who Masked: Participant, Care Provider
Masking Description: Model Description Model Description Definition: Provide details about the Interventional Study Model. Limit: 1000 characters.Model Description Definition: Provide details about the Interventional Study Model. Limit: 1000 characters.Model Description Definition: Provide details about the Interventional Study Model. Limit: 1000 characters.Model Description Definition: Provide details about the Interventional Study Model. Limit: 1000 characters.Model Description Definition: Provide details about the Interventional Study Model. Limit: 1000 characters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P3-T PrEP adherence app (Experimental): Intended app use includes, at a minimum, participant completion of selected app activities (medication tracking, daily quest, social wall post) each day for the 3 month intervention period.
  Participant completion of Standard of Care PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and the 4-month post-prescription visit.
  Interventions: Behavioral: P3-T PrEP Adherence App
- Standard of Care (No Intervention): Participant completion of Standard of Care PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and the 4-month post-prescription visit.

INTERVENTIONS:
Behavioral: P3-T PrEP Adherence App — P3-T provides daily PrEP reminders, a medication tracker and calendar, personalized medication adherence strategies, refill reminders, and tailored adherence support messages; social support via a social wall that includes daily discussion prompts; daily quests to build knowledge and skills; a multimedia knowledge center; interactive narrative collections; personalized adherence counseling provided by an adherence counselor via in-app messaging; in-app rewards; a "bank account" that rewards daily app use by adding or subtracting a small financial reward based on daily app use; and, a user profile that includes a user-selected avatar.
  Other Names: P3-T
  Arms: P3-T PrEP adherence app

SUMMARY:
This study aims to: 1) adapt the theory-based P3 (Prepared, Protected, emPowered) app designed to improve pre-exposure prophylaxis (PrEP) adherence, retention in PrEP clinical care, and PrEP persistence among young gay, bisexual, and other men who have sex with men (YMSM) in the United States for YMSM in Thailand, and 2) conduct a pilot randomized controlled trial (RCT) to assess the feasibility, acceptability, and potential impact of the adapted P3-Thailand (P3-T) app.

DETAILED DESCRIPTION:
This R21 study, titled "Novel mHealth Technologies to Enhance PrEP Adherence among Thai MSM: Collaborative Adaptation and Evaluation" was designed to adapt and test a theory-based, PrEP adherence smartphone app, P3, to 1) improve PrEP adherence and thus protective PrEP drug levels, 2) to increase retention in PrEP clinical care, 3) support PrEP persistence among YMSM in the United States for YMSM in Thailand, and 4) conduct a pilot RCT to assess the feasibility and acceptability of the adapted P3-T app and to examine the potential impact of the app on PrEP adherence.

The study was a partnership between Duke University, Chulalongkorn University, Thai Red Cross AIDS Research Centre (TRC-ARC), and the University of North Carolina-Chapel Hill, and includes a robust plan to increase mHealth capacity at Chulalongkorn University and TRC-ARC.

P3 is a theory-based, comprehensive smartphone app platform for YMSM that utilizes social networking and game-based mechanics as well as evidenced-based features to improve PrEP medication adherence. P3 is a product born from the collaborative effort of researchers and health game developers working closely with members of the target population in the United States. Built on a successful, evidence-based platform designed by our collaborating technology partner, Ayogo, and tested by our study team, P3 is flexible, allowing for customization and adaptations for different cultural and linguistic contexts, and responsive to changes in technology.

The social networking features of P3 are designed to capitalize on social involvement as a means through which YMSM can receive information and social support, experience social norms and reflective appraisals, and feel a sense of connectedness to peers. Peers have been recognized as a highly important source of sexual health and HIV prevention information and support among Thai YMSM. The gaming features of P3 were goal-oriented and immersive and provided a challenging and motivating environment for behavior change. As a result, P3 is ideal for engaging YMSM in behavior change, by maintaining attention and avoiding boredom and attrition.

The pilot RCT of the adapted P3-T app was conducted with 60 YMSM newly starting PrEP in Bangkok, Thailand to 1) assess app feasibility and acceptability, and 2) explore the potential impact of the app on PrEP adherence.

In-depth interviews were conducted with 10 P3-T arm participants after the 3-month intervention period. The interview will ask participants about their experience and impressions of the app, how they used it, and how it may have impacted their behaviors during the 3-month intervention period.

ELIGIBILITY:
Inclusion Criteria

* Male sex at birth
* Gender identity is male
* Identify as a man who has sex with men
* Ages 16-24
* Plan to start PrEP in next 14 days
* Able to speak and read Thai
* Own an Android or iOS smartphone

Exclusion Criteria:

* Currently participating in another experimental PrEP adherence intervention
* Plan to move out of Bangkok in the next 6 months
* Unable to be consented due to an active substance use or psychological condition

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-identify as male
Enrollment: 60 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara LeGrand, Ph.D., Principal Investigator — Duke University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Songtaweesin WN, LeGrand S, Bandara S, Piccone C, Wongharn P, Moonwong J, Jupimai T, Saisaengjan C, Theerawit T, Muessig K, Hightow-Weidman L, Puthanakit T, Phanuphak N, Tangmunkongvorakul A. Adaptation of a Theory-Based Social Networking and Gamified App-Based Intervention to Improve Pre-Exposure Prophylaxis Adherence Among Young Men Who Have Sex With Men in Bangkok, Thailand: Qualitative Study. J Med Internet Res. 2021 Nov 4;23(11):e23852. doi: 10.2196/23852. PMID 34734828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited by study staff based on physician referral to the Chulalongkorn pre-exposure prophylaxis (PrEP) clinic in Bangkok, Thailand between June 12, 2020 and January 15, 2021.
Pre-assignment Details: 60 individuals met the study inclusion criteria and were enrolled and randomized into the P3T arm or the Standard of Care arm.
Groups:
- P3-T PrEP Adherence App: P3-T provided daily PrEP reminders, a medication tracker and calendar, personalized medication adherence strategies, refill reminders, and tailored adherence support messages; social support via a social wall that included daily discussion prompts; daily quests to build knowledge and skills; a multimedia knowledge center; interactive narrative collections; personalized adherence counseling provided by an adherence counselor via in-app messaging; in-app rewards; a "bank account" that rewards daily app use by adding or subtracting a small financial reward based on daily app use; and, a user profile that included a user-selected avatar.
  Intended app use includes, at a minimum, participant completion of selected app activities (medication tracking, daily quest, social wall post) each day for the 3-month intervention period.
  Participant completion of Standard of Care PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and the 4-month post-prescription visit.
  Other Name: P3-T
Period: Overall Study
Arm/Group | P3-T PrEP Adherence App | Standard of Care
Started | 30 | 30
Completed | 29 | 28
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: The primary analysis population included young, gay, bisexual, and other men who have sex with men, ages 16-24, who were initiating preexposure prophylaxis (PrEP). Individuals were randomized 1:1 into either the P3-T app intervention + standard of care or the standard of care arm. Study participants completed a Qualtrics survey at baseline, M3, and M6. At M3 and M6 dried blood spots were collected for tenofovir diphosphate (TFV-DP) to quantify PrEP adherence levels.
Groups:
- P3-T PrEP Adherence App: Intended app use includes, at a minimum, participant completion of selected app activities (medication tracking, daily quest, social wall post) each day for the 3 month intervention period.
  Participant completion of Standard of Care PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and the 4-month post-prescription visit.
  P3-T PrEP Adherence App: P3-T provides daily PrEP reminders, a medication tracker and calendar, personalized medication adherence strategies, refill reminders, and tailored adherence support messages; social support via a social wall that includes daily discussion prompts; daily quests to build knowledge and skills; a multimedia knowledge center; interactive narrative collections; personalized adherence counseling provided by an adherence counselor via in-app messaging; in-app rewards; a "bank account" that rewards daily app use by adding or subtracting a small financial reward based on daily app use; and, a user profile that includes a user-selected avatar.
- Total: Total of all reporting groups
Arm/Group | P3-T PrEP Adherence App | Standard of Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21 [20 to 21] | 22 [20 to 23] | 21 [20 to 22]
Sex/Gender, Customized [Number; unit: participants]
  Assigned male sex at birth | 30 | 30 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 30 | 30 | 60
Current sexual identity [Count of Participants; unit: Participants]
  Gay, homosexual, same gender loving | 22 | 24 | 46
  Bisexual | 5 | 3 | 8
  Queer | 2 | 2 | 4
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility: Average Number of Days of Any App Use
Description: The number of days of any app use among those assigned to the P3-T adherence arm during the 3-month intervention period as recorded by backend app metrics. Higher number of days indicates higher intervention feasibility.
Time Frame: Month 3
Population: Only applies to P3-T PrEP Adherence App group
Measure: Mean (Standard Deviation); unit: days
Arm/Group | P3-T PrEP Adherence App
Number analyzed (Participants) | 30
days | 68 (29)

2. Primary Outcome: Intervention Feasibility: Average Number of Days of PrEP Medication Tracked Through App
Description: The number of days of PrEP medication tracked through app during the 3-month intervention period among participants assigned to the P3-T adherence arm as recorded by backend app metrics. Higher number indicates higher intervention feasibility.
Time Frame: Month 3
Population: Only applies to P3-T PrEP Adherence App group
Measure: Mean (Standard Deviation); unit: Days
Groups:
- P3-T PrEP Adherence App: Intended app use includes, at a minimum, participant completion of selected app activities (medication tracking, daily quest, social wall post) each day for the 3-month intervention period. Participant completion of Standard of Care PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and the 4-month post-prescription visit.
  P3-T PrEP Adherence App: P3-T provides daily PrEP reminders, a medication tracker and calendar, personalized medication adherence strategies, refill reminders, and tailored adherence support messages; social support via a social wall that includes daily discussion prompts; daily quests to build knowledge and skills; a multimedia knowledge center; interactive narrative collections; personalized adherence counseling provided by an adherence counselor via in-app messaging; in-app rewards; a "bank account" that rewards daily app use by adding or subtracting a small financial reward based on daily app use; and, a user profile that includes a user-selected avatar.
Arm/Group | P3-T PrEP Adherence App
Number analyzed (Participants) | 30
Days | 60 (28)

3. Primary Outcome: Intervention Acceptability: Mean Intervention Acceptability, Composite Score CSQ-8
Description: Intervention acceptability was assessed using the Client Satisfaction Questionnaire (CSQ-8), an 8-item validated scale measuring the construct of global intervention satisfaction, collected in the 3-month follow-up survey (intervention group only). The eight items (quality of app, kind of service received from app, app met needs, recommend app to a friend, amount of help received from app, the effectiveness of app for dealing with health issue (PrEP adherence), overall satisfaction, and willingness to use the app again) were assessed using a 4-point response scale with individually specified anchors. The mean composite score of the CSQ-8 was calculated with a total possible range of 8 (lowest acceptability, worst outcome) to 32 (highest acceptability, best outcome).
Time Frame: Month 3
Population: Only applies to P3-T PrEP Adherence App group. Data not collected on 2 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- P3-T PrEP Adherence App: P3-T provided daily PrEP reminders, a medication tracker and calendar, personalized medication adherence strategies, refill reminders, and tailored adherence support messages; social support via a social wall that included daily discussion prompts; daily quests to build knowledge and skills; a multimedia knowledge center; interactive narrative collections; personalized adherence counseling provided by an adherence counselor via in-app messaging; in-app rewards; a "bank account" that rewards daily app use by adding or subtracting a small financial reward based on daily app use; and, a user profile that included a user-selected avatar.Intended app use includes, at a minimum, participant completion of selected app activities (medication tracking, daily quest, social wall post) each day for the 3-month intervention period.
  Participant completion of Standard of Care PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and the 4-month post-prescription visit.
Arm/Group | P3-T PrEP Adherence App
Number analyzed (Participants) | 28
score on a scale | 25.18 (4.11)

4. Secondary Outcome: Difference in PrEP Medication Adherence Between Study Arms at Month 3
Description: The number of participants with protective levels of tenofovir-diphosphate (TFV-DP) at month 3 between the study arms.
Time Frame: Month 3
Population: Data not collected on 4 participants.
Measure: Number; unit: count of participants
Groups:
- P3-T PrEP Adherence App: P3-T provided daily PrEP reminders, a medication tracker and calendar, personalized medication adherence strategies, refill reminders, and tailored adherence support messages; social support via a social wall that included daily discussion prompts; daily quests to build knowledge and skills; a multimedia knowledge center; interactive narrative collections; personalized adherence counseling provided by an adherence counselor via in-app messaging; in-app rewards; a "bank account" that rewards daily app use by adding or subtracting a small financial reward based on daily app use; and, a user profile that included a user-selected avatar.
  Intended app use includes, at a minimum, participant completion of selected app activities (medication tracking, daily quest, social wall post) each day for the 3-month intervention period.
  Participant completion of Standard of Care PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and the 4-month post-prescription visit.
Arm/Group | P3-T PrEP Adherence App | Standard of Care
Number analyzed (Participants) | 29 | 27
count of participants | 27 | 23
Statistical Analysis 1: Comparison: P3-T PrEP Adherence App vs Standard of Care; Test type: Superiority; p = 0.41, Fisher Exact; Risk Ratio (RR) = 1.62, 95% CI 2-sided [0.50 to 5.17]

5. Secondary Outcome: Difference in PrEP Medication Adherence Between Study Arms at Month 6
Description: The number of participants with protective levels of TFV-DP at month 6 between the study arms.
Time Frame: Month 6
Population: Data not collected on 5 participants
Measure: Count of Participants; unit: Participants
Arm/Group | P3-T PrEP Adherence App | Standard of Care
Number analyzed (Participants) | 29 | 26
Participants | 21 | 18
Statistical Analysis 1: Comparison: P3-T PrEP Adherence App vs Standard of Care; Test type: Superiority; p = 1.0, Fisher Exact; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.61 to 1.90]

ADVERSE EVENTS:
Time Frame: Approximately 6 months
Groups:
- P3-T PrEP Adherence App: P3-T provided daily PrEP reminders, a medication tracker and calendar, personalized medication adherence strategies, refill reminders, and tailored adherence support messages; social support via a social wall that included daily discussion prompts; daily quests to build knowledge and skills; a multimedia knowledge center; interactive narrative collections; personalized adherence counseling provided by an adherence counselor via in-app messaging; in-app rewards; a "bank account" that rewards daily app use by adding or subtracting a small financial reward based on daily app use; and, a user profile that included a user-selected avatar. Intended app use included, at a minimum, participant completion of selected app activities (medication tracking, daily quest, social wall post) each day for the 3-month intervention period.
  Participant completion of Standard of Care PrEP adherence and sexual risk behavior counseling at the 1-month post-prescription visit and the 4-month post-prescription visit.
Arm/Group | P3-T PrEP Adherence App | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT04413708/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT04413708/ICF_001.pdf